CLINICAL TRIAL: NCT01162707
Title: A Multi-Center, Non-Randomized, Prospective Trial to Evaluate the Safety and Feasibility of Wireless, Intermittent Monitoring of Right Heart Pressures in Adult Heart Failure Subjects
Brief Title: Wireless, Intermittent Monitoring of Right Heart Pressures in HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CardioMEMS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM-06-03
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: NYHA Class III Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pressure Measurement System (Experimental): CardioMEMS HF Pressure Measurement System
  Interventions: Device: CardioMEMS HF Pressure Measurement System

INTERVENTIONS:
Device: CardioMEMS HF Pressure Measurement System — Implant sensor into the left or right pulmonary artery. Measure pulmonary artery pressure

SUMMARY:
The purpose of the trial is to evaluate the wireless monitoring of pulmonary artery pressure using the CardioMEMS HF Pressure Measurement System in adult subjects with NYHA Class III Heart Failure.

DETAILED DESCRIPTION:
The trial is designed to demonstrate that the CardioMEMS Sensor can be positioned in the right or left pulmonary artery, and that Sensor pressure measurements correlate to standardized methods of intra-cardiac pressure measurements post-sensor implant and at the 60 day visit. Safety will be monitored by the occurrence of adverse events throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, at least 18 years of age
2. Subjects of childbearing age who have a negative serum pregnancy test, and at screening have agreed to use a reliable mechanical or hormonal form of conception during the study.
3. Subject has a diagnosis of New York Heart Association (NYHA) Class III HF at screening and at baseline.
4. Subject is able and willing to provide written informed consent or the subject guardian is able and willing to provide informed consent.
5. Subject has life expectancy of 1-2 years.

Exclusion Criteria:

1. Subject has unstable medical condition or impairment other than a medical condition associated with HF which would significantly increase the subject's morbidity or mortality risk.
2. Subject is unable to tolerate a right heart catheterization.
3. Subject is planned to undergo a heart transplantation or cardiac surgery within 2 months after enrollment.
4. Subject has permanent indwelling central venous catheter.
5. Subject has history of myocardial infarction (MI), unstable angina, stroke, transient ischemic attack, or intractable arrhythmias within last 2 months.
6. Subject has history of congenital heart disease or prosthetic valve on right side.
7. Subject has unstable hypertension.
8. Subject has a known coagulability disease state.
9. Subject has a known hypersensitivity and/or allergy to aspirin and clopidogrel.
10. Subject has active lung infection or acute pulmonary decompensation.
11. Subject has elevated white blood cell count and signs of infection are evident.
12. Subject has chronic renal insufficiency as defined by serum creatinine of greater than or equal to 2 mg/dl or requirement for dialysis.
13. Subject who is pregnant or lactating or might become pregnant during the duration of the study.
14. Subject who is participating in another therapeutic interventional trial.
15. Subject has other medical, psychological, or social circumstances that may affect the ability to comply with the study requirements or increase risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-12; Primary Completion 2007-11 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the wireless monitoring of pulmonary artery pressure using the CardioMEMS HF Pressure Measurement System in adult subjects with Class III Heart Failure. | after implant of the sensor and at 60 day visit
  The trial will demonstrate that the CardioMEMS Sensor can be positioned in the right or left pulmonary artery, and the Sensor pulmonary artery pressure measurements correlate to standardized methods of intra-cardiac pressure measurements immediately after deployment of the sensor and at the 60 day follow-up visit. Safety is assessed by monitoring the occurrence of adverse events.

SECONDARY OUTCOMES:
To demonstrate the capability of the CardioMEMS HF System to obtain the pressure measurement from the Sensor and transmit the pulmonary artery pressure data to a secure database. | after deployment of the sensor and at 60 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Piedmont Hospital, Atlanta, Georgia
  - Ohio State University Hospital, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - St Thomas Hospital, Nashville, Tennessee